CLINICAL TRIAL: NCT06995612
Title: SMART-CPT for PTSD and History of Concussion: A Pragmatic Implementation Trial
Brief Title: SMART-CPT for PTSD/Concussion Implementation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy Jak, Principal Investigator, San Diego Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP220123
Record Dates: First submitted 2024-01-05; First posted 2025-05-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-03

CONDITIONS: PTSD; Concussion, Mild
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Concussion | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMART-CPT (Experimental)
  Interventions: Behavioral: SMART-CPT
- CPT (Active Comparator)
  Interventions: Behavioral: CPT

INTERVENTIONS:
Behavioral: SMART-CPT — SMART-CPT T is a psychotherapy that combines Cognitive Processing Therapy (CPT) for Posttraumatic Stress Disorder (PTSD) and Cognitive Symptom Management and Rehabilitation Training (CogSMART) for neurobehavioral and neurocognitive symptoms to simultaneously target persistent postconcussive symptoms and PTSD
  Arms: SMART-CPT
Behavioral: CPT — CPT is a cognitive behavioral treatment specifically targeting PTSD and other corollary symptoms following traumatic events (Resick & Schnicke, 1992). Based on a social cognitive theory of PTSD and trauma, CPT focuses on identifying the content of trauma-related thoughts, examining whether these thoughts are consistent or inconsistent with a patient's prior beliefs about the world, and addressing the impact these thoughts have on emotions and behaviors. Patients are taught to recognize and challenge thought patterns such as, assimilation (distorting the memory of the traumatic event to fit prior world beliefs), over-accommodation (excessively altering world beliefs to be consistent with the trauma), or the reinforcement of previously held distorted world beliefs.
  Arms: CPT

SUMMARY:
The clinical implementation trial will evaluate effectiveness and feasibility, acceptability, appropriateness, barriers, and facilitators of implementing SMART-CPT, a treatment targeting the two primary factors leading to poor outcomes following concussion, in Veterans. It will test effectiveness and broad implementation feasibility of SMART-CPT compared to standard Cognitive Processing Therapy (CPT).

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis;
* mild TBI sustained greater than three months prior to enrollment;
* cognitive complaints;
* not medicated or stable on prescribed psychiatric medication for at least 6 weeks prior to study enrollment with no anticipated/pending medication changes;
* English literacy.

Exclusion Criteria:

* mTBI sustained less than 3 months previously;
* history of moderate, severe, or penetrating TBI;
* history of other significant neurological condition unrelated to TBI;
* severe psychiatric disturbance expected to interfere with successful completion of the study;
* current severe alcohol or other substance use disorder;
* suicidal intent or attempt within the previous month;
* current homicidal ideation;
* impaired decision making capacity;
* prior completion of five or more sessions of CPT or cognitive rehabilitation; -concurrent participation in other intervention studies for PTSD or TBI;
* life threatening or unstable medical illness;
* inability to read;
* dementia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist (PCL5) | weekly through treatment completion, an average of 3 months
  A brief self-report instrument to measure PTSD symptom severity. It consists of 20 items, scored on a 5-point scale (0 = not at all to 5 = extremely), that correspond to the DSM-5 symptoms of PTSD. It will be used to track PTSD symptom reporting weekly as well as at comprehensive assessments
Neurobehavioral Symptom Inventory (NSI) | weekly through treatment completion, an average of 3 months
  A 22 item self-report measure of neurobehavioral symptoms commonly experienced following a mTBI that will be utilized to assess inclusionary cognitive complaints as well as monitor overall neurobehavioral symptoms weekly and at comprehensive assessments.
The Patient Global Impression of Change (PGIC) | at treatment completion, an average of three months
  A single-item measure of activity limitations, symptoms, and overall quality of life
Brief Inventory of Psychosocial Functioning (B-IPF) | at 3 primary assessment timepoints, week 0, week 12, week 24
  7-item measure of PTSD psychosocial functional impairment
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | at 3 primary assessment timepoints; week 0, week 12, week 24
  will measure function in the following areas: life activities (work, school, domestic responsibilities), cognition, mobility, self-care, social, and community participation
Traumatic Brain Injury Quality of Life Scale (TBI-QOL) | at 3 primary assessment timepoints; week 0, week 12, week 24
  provides comprehensive patient-reported outcomes specific to TBI.

CONTACTS AND LOCATIONS:
Locations (1):
- VA San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be uploaded to FITBIR for aggregation and secondary analyses by other investigators.
Supporting Information: Study Protocol
Time Frame: at study completion
Access Criteria: FITBIR is publicly available researchers at fitbir.nih.gov
URL: http://fitbir.nih.gov